CLINICAL TRIAL: NCT01555450
Title: The Patient Navigator to Reduce Social Inequalities. A French Interventional Trial in Public Health
Brief Title: Study of Patient Navigation to Reduce Social Inequalities
Acronym: PRADO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: R10051EE
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2012-03

CONDITIONS: Colorectal Cancer Screening
Keywords: Colorectal cancer screening; Social inequalities; Patient Navigator
MeSH Terms: interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- With Patient Navigator (Experimental): People in this arm receive the Intervention of a Patient Navigator
  Interventions: Other: Patient Navigation
- Control - Without Patient Navigator (No Intervention): People in this arm receive just the usual care of colorectal cancer screening

INTERVENTIONS:
Other: Patient Navigation — Insured people receive firstly a letter to inform them that a patient navigator is available to navigate them during the colorectal screening steps. A free telephone number and the navigator schedule is given. After a minimum of one week the patient navigator begins the telephone outreach.
  Arms: With Patient Navigator

SUMMARY:
Variations in participation to the colorectal cancer screening seems to reveal social and geographical inequalities. Our study will investigate whether patient navigation could increase the participation to the colorectal cancer screening and in the same time, reduce the social inequalities.

ELIGIBILITY:
Inclusion Criteria:

* Insured people invited to the national french colorectal screening program are from 50 to 74 years old.
* We select people who never do the screening test or are not compliant with it
* Among these people we select those living in the randomized geographical areas.

Exclusion Criteria:

* people who have already done the screening test at the two previous campaigns.
* people who have done a colonoscopy in the previous five years or people with a family history with colorectal cancer and people who are following outside of the screening program.
* people with other severe disease or in incapacity to realize the screening test
* people who have another exclusion criteria to realize the screening test.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28929 (Actual)
Dates: Start 2011-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Completion of colorectal cancer screening | 2 years
Reduction of social inequalities | 2 years
  The participation rate to the colorectal cancer screening will be compared between privileged and deprived geographical areas for which the socio-economic status is measured with the Townsend index.

SECONDARY OUTCOMES:
Estimation of Cost effectiveness | 2 years
  We will assess the mean cost to navigate one person and compared it to a non navigate person. We will measure the cost effectiveness of the intervention in order to have the cost of the arising of 1% of the participation rate.
Evaluation of psychological mechanisms | 2 years
  Evaluation of cognitive, behavioural, emotional mechanisms influencing the colorectal screening participation

CONTACTS AND LOCATIONS:
Overall Officials: Guy Launoy, Pr, Study Director — CHU CAEN / INSERM
Locations (3):
- France (3):
  - The french screening organization, Amiens, Region of Picardie
  - The french screening organization, Compiègne, Region of Picardie
  - The french screening organization, Laon, Region of Picardie

REFERENCES:
- [Background] Dejardin O, Berchi C, Mignon A, Pornet C, Guillaume E, Guittet L, Bouvier V, Sailly M, Salinas A, Christophe V, Launoy G. [Social inequalities in health from observational studies to intervention: can the patient navigator reduce social inequalities in cancer patients?]. Rev Epidemiol Sante Publique. 2011 Feb;59(1):45-51. doi: 10.1016/j.respe.2010.10.008. Epub 2011 Jan 21. French. PMID 21256688
- [Result] De Mil R, Guillaume E, Guittet L, Dejardin O, Bouvier V, Pornet C, Christophe V, Notari A, Delattre-Massy H, De Seze C, Peng J, Launoy G, Berchi C. Cost-Effectiveness Analysis of a Navigation Program for Colorectal Cancer Screening to Reduce Social Health Inequalities: A French Cluster Randomized Controlled Trial. Value Health. 2018 Jun;21(6):685-691. doi: 10.1016/j.jval.2017.09.020. Epub 2017 Nov 10. PMID 29909873
- [Result] Guillaume E, Dejardin O, Bouvier V, De Mil R, Berchi C, Pornet C, Christophe V, Notari A, Delattre Massy H, De Seze C, Peng J, Guittet L, Launoy G. Patient navigation to reduce social inequalities in colorectal cancer screening participation: A cluster randomized controlled trial. Prev Med. 2017 Oct;103:76-83. doi: 10.1016/j.ypmed.2017.08.012. Epub 2017 Aug 16. PMID 28823681